CLINICAL TRIAL: NCT06580028
Title: Electroencephalogram Study in Children Under Sevoflurane Anesthesia - a Prospective,Observational Study
Brief Title: The EEG Study Under Sevoflurane Anesthesia in Children
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-03-217
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Electroencephalography; Sevoflurane; Child Neglect
Keywords: Sevoflurane; Children; Electroencephalogram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- 0-3 months: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 3-6 months: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 6-9 months: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 9-12 months: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 1-1.5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 1.5-2 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 2-2.5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 2.5-3 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 3-3.5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 3.5-4 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 4-4.5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 4.5-5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 5-5.5 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.
- 5.5-6 years: EEG was collected during the whole perioperative period, including preoperative conscious period (or preoperative sedation period) , anesthesia period and anesthesia recovery period.

SUMMARY:
Sevoflurane is one of the most commonly used volatile anesthetics in children because of its rapid induction, recovery and recovery properties. Clinical studies using noninvasive brain monitoring have shown that general anesthetics and hypnotics generate electroencephalogram (EEG) oscillations in specific spatial tissues that are fundamentally related to the structure and function of neural circuits. Slow-wave-delta (0.1-4 Hz) oscillations were present in children of all ages, and the advantage of frontal α-wave oscillations appeared at approximately 6 months, began to be consistent at 10 months, and persisted at older ages. Another study, which analyzed EEG under sevoflurane general anesthesia in children aged 0-6 months, found that Theta and alpha wave power decreased with a decrease in sevoflurane concentrations in infants between 4 and 6 months of recovery. However, these studies lack detailed characterization of the neural circuit activity associated with anesthesia, especially at specific developmental ages that are highly correlated with brain plasticity. The aim of this study was to explore electroencephalogram (EEG) of children of different ages under sevoflurane general anesthesia (including anesthesia induction, maintenance and recovery) . By analyzing these EEG data in detail, we hope to be able to better understand the EEG characteristics of children of different ages under sevoflurane anesthesia, and thus develop a neurophysiology pediatric anesthesia status monitoring strategy.

DETAILED DESCRIPTION:
This study is prospective and observational. Children under sevoflurane general anesthesia were divided into 14 groups (0-3 months old, 3-6 months old, 6-9 months old, 9-12 months old, 1-1.5 years old, 1.5-2 years old, 2-2.5 years old, 2.5-3 years old, 3-3.5 years old, 3.5-4 years old, 4-4.5 years old, 4.5.5 years old, 5.5.5 years old, 5.5-6 years old) , there were 20 cases in each group. Inform the family about the research plan and obtain informed consent. To observe the time-frequency characteristics of prefrontal electroencephalogram (EEG) in children of different ages under general anesthesia with sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

1. aged 1 days#6 years#;
2. with American Society of Anesthesiologists (ASA) physical status I or II#;
3. children requiring general anesthesia under sevoflurane;
4. parents or legal guardians of children who volunteered to participate in the trial; And signed the informed consent form.

Exclusion Criteria:

1. Congenital malformation or other genetic conditions that are thought to affect brain development ;
2. History of severe heart, brain, liver, kidney and metabolic diseases ;
3. Premature infants (≤32 weeks);
4. Upper respiratory tract infection in the last two weeks.

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population met the above inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Time-frequency characteristics of electroencephalogram (EEG) | during sevoflurane general anesthesia (including anesthesia induction, maintenance and recovery)
  Time-frequency characteristics of electroencephalogram (EEG) in children of different ages during sevoflurane general anesthesia (including anesthesia induction, maintenance and recovery) .

SECONDARY OUTCOMES:
Modified observer's assessment of alertness#sedation#MOAA/S#scale | during sevoflurane general anesthesia (including anesthesia induction, maintenance and recovery)
  5#Subject responds readily to name spoken in a normal tone; 4 #Lethargic response of a subject to a name spoken in a normal tone; 3 #The subject responds only after a name is called loudly and repeatedly; 2 #The subject responds only after mild prodding or shaking;
  1 #The subject responds only after a painful trapezius squeeze; 0 #The subject does not respond to painful trapezius squeeze. MOAA/S score ≤ 2 points represent successful sedation
Recovery time | Within up to 30 minutes after operation
  From the time sevoflurane was stopped until the child opened his eyes for the first time and reached an Aldrete score of ≥9
Pediatric anesthesia emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
The Face, Legs, Activity, Cry, Consolability Scale (FLACC) | Within up to 30 minutes after operation
  The FLACC scale consists of five items. Each item is scored 0-2 yielding a total between 0 and 10.
PHBQ-AS | 3 days after operation
  Post-Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS) is a parental report measure used to assess negative behavior change after hospitalization, consisting of 11 items on 1-5 score. The PHBQ-AS score will be calculated for each respondent as the mean score of all individual items answered on the questionnaire.
  A score above 3 will indicate the presence of negative behavioral change, a score equal to 3 will indicate no behavioral change, and a score below 3 will indicate an improvement in behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China